CLINICAL TRIAL: NCT01767428
Title: A Pharmacokinetic Study to Evaluate the Rate and Extent of Absorption of Paracetamol From Two Formulations in an Indian Population.
Brief Title: Pharmacokinetic Study to Compare Two Formulations of Paracetamol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A1900832
Record Dates: First submitted 2012-12-06; First posted 2013-01-14 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Fever; Headache Disorders; Pain
MeSH Terms: conditions — Fever; Headache Disorders; Pain | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Paracetamol Tablet (Experimental): Experimental paracetamol tablet (500 milligrams [mg]) administered with 240 milliliters (mL) of water.
  Interventions: Drug: Paracetamol
- Standard Paracetamol Tablet (500 mg) (Active Comparator): Standard paracetamol tablet (500 mg) administered with 240 mL of water.
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — 500 mg immediate release paracetamol formulations

SUMMARY:
A pharmacokinetic study in healthy volunteers comparing two formulations of paracetamol fast release in fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18-55yrs willing to give written informed consent for the study
* BMI must be within the range 18.5 - 24.9 kg/m^2
* Participant with a minimum weight of 50 kg

Exclusion Criteria:

* Participant with current or recurrent disease that could affect the action, absorption or disposition of the study medication or clinical or laboratory assessments (e.g. hepatic disorders, renal insufficiency, congestive heart failure)
* Participant with known or suspected intolerance or hypersensitivity to the study materials
* Participant who are vegetarian
* Participant smoking more than five cigarettes a day

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
AUC (0-inf) | Blood samples drawn at 15 minutes pre-dose, then at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 60, 75, 90 minutes post dose and then at 2, 3, 4, 6, 8, 10, 12 hrs post dose.
  Area under the plasma concentration time curve from zero and extrapolated to infinite time.
Cmax | Blood samples drawn at 15 minutes pre-dose, then at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 60, 75, 90 minutes post dose and then at 2, 3, 4, 6, 8, 10, 12 hrs post dose.
  Maximum plasma concentration of paracetamol.
AUC (0-t) | Blood samples drawn at 15 minutes pre-dose, then at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 60, 75, 90 minutes post dose and then at 2, 3, 4, 6, 8, 10, 12 hrs post dose.
  Area under the plasma concentration time curve from zero and extrapolated to the time of last quantifiable sample.

SECONDARY OUTCOMES:
Tmax | Blood samples drawn at 15 minutes pre-dose, then at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 60, 75, 90 minutes post dose and then at 2, 3, 4, 6, 8, 10, 12 hrs post dose.
  Time taken to reach maximum plasma concentration of paracetamol.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline